CLINICAL TRIAL: NCT06277024
Title: A Study on the Safety and Efficacy of the Combination of Candenizumab, Lenvatinib, and SOX Regimen in the Treatment of HER2 Negative Advanced Gastric or Gastroesophageal Junction Adenocarcinoma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., chief physician, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-32
Record Dates: First submitted 2024-02-04; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Overall Response Rate
Keywords: gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with combination of candenizumab, lenvatinib, and SOX regimen (Experimental)
  Interventions: Drug: Combination of Cardonizumab with Lenvatinib and SOX regimen

INTERVENTIONS:
Drug: Combination of Cardonizumab with Lenvatinib and SOX regimen — Phase 1: Conduct a ramp up test on the dosage of lenvatinib according to the traditional 3+3 design; Phase 2: 6 cycles of treatment with candenizumab+lenvatinib+SOX regimen (Q3W); For patients who have not progressed, they will enter the third stage of maintenance treatment.
  Phase 3: Maintenance therapy with candenizumab, lenvatinib, and tigio (Q3W).

SUMMARY:
Evaluate the objective response rate (ORR) of the combination of candenizumab, lenvatinib, and SOX regimen for the treatment of HER2 negative advanced gastric or gastroesophageal junction adenocarcinoma patients

DETAILED DESCRIPTION:
Local advanced or metastatic HER2 negative gastric or gastroesophageal junction adenocarcinoma confirmed by histopathology or cytology that cannot be resected, and has not received systemic treatment (including HER2 inhibitors) as the primary treatment for advanced or metastatic diseases in the past.

Evaluate the objective response rate (ORR) of the combination of candenizumab, lenvatinib, and SOX regimen for the treatment of HER2 negative advanced gastric or gastroesophageal junction adenocarcinoma patients Median survival time (OS);

* Progression free survival time (PFS);
* Duration of relief (DOR); Evaluate the safety of this regimen in the treatment of advanced gastric or gastroesophageal junction adenocarcinoma patients, including the incidence of adverse events (AE), severe adverse reactions (SAE), dose adjustment rate, and dose pause rate; Observe the changes in quality of life of patients with advanced gastric or gastroesophageal junction adenocarcinoma after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years ≤ Age ≤ 75 years;
* Locally advanced or metastatic HER2 negative gastric or gastroesophageal junction adenocarcinoma confirmed by histopathology or cytology that cannot be resected;
* Has not received radiotherapy, chemotherapy, targeted therapy, or immunotherapy as the primary treatment option for advanced or metastatic diseases in the past; Participants with gastric or gastroesophageal junction adenocarcinoma who have previously received adjuvant or neoadjuvant chemotherapy, radiotherapy, and/or radiochemotherapy are eligible for enrollment as long as the last administration of the previous protocol occurred at least 6 months prior to randomization.
* At least one measurable lesion #see Appendix 2#;
* ECOG PS: 0-1 points #see Appendix 4#;
* Estimated survival time>3 months;
* The main organ function is normal and meets the following criteria:
* Blood routine examination must meet the following criteria#no blood transfusion within 14 days#

  1. HB ≥ 100g/L,
  2. WBC ≥ 3 × 109/L
  3. ANC ≥ 1.5 × 109/L,
  4. PLT ≥ 100 × 109/L;
* Biochemical examination must meet the following standards:

  1. BIL<1.5 times the upper limit of normal value #ULN#,
  2. ALT and AST<2.5ULN, GPT ≤ 1.5 × ULN;
  3. Serum Cr ≤ 1ULN, endogenous creatinine clearance rate>60ml/min #Cockcroft Gault formula#
* Women of childbearing age must undergo a pregnancy test #serum# within 7 days before enrollment, and the result is negative. They are willing to use appropriate methods of contraception during the trial period and 8 weeks after the last administration of the trial drug; For males, surgical sterilization or agreement to use appropriate methods of contraception during the trial period and 8 weeks after the last administration of the trial drug should be considered; 9# Not participating in other clinical studies before and during treatment; 10# The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* If a subject meets any of the following conditions, they will not be allowed to enter this study

  * Patients with allergies or suspected allergies to research drugs or similar drugs;
  * Suffering from other malignant tumors within the past 5 years, excluding skin basal cell or squamous cell carcinoma after radical surgery, or cervical carcinoma in situ;
  * Received live vaccine within 4 weeks prior to enrollment or possibly during the study period;
  * Suffering from active autoimmune diseases or having a history of autoimmune diseases within 4 weeks prior to enrollment;
  * Previously received allogeneic bone marrow transplantation or organ transplantation;
  * The patient currently has any disease or condition that affects drug absorption, or the patient is unable to take medication orally;
  * The patient currently has hypertension that cannot be controlled by medication, which is defined as: patients with hypertension who cannot be well controlled with a single antihypertensive drug treatment #systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100mmHg#; Or use two or more antihypertensive drugs to control blood pressure in patients;
  * Urinary routine indicates that urine protein is ≥ 2+, and the 24-hour urine protein volume is>1.0g;
  * The patient currently has digestive tract diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresectable tumors, or other conditions determined by the researcher that may cause gastrointestinal bleeding or perforation;
  * Patients with significant evidence of bleeding tendency or medical history within the 3 months prior to enrollment #bleeding>30 mL within 3 months, vomiting blood, black stool, and rectal bleeding#, hemoptysis #fresh blood>5 mL within 4 weeks#, or thromboembolic events #including stroke events and/or transient ischemic attacks# within 12 months;
  * Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting surgery within 6 months prior to enrollment; Congestive heart failure is classified by the New York Heart Association #NYHA# as>level 2; Ventricular arrhythmia requiring medication treatment; Electrocardiogram #ECG# shows a QT interval of ≥ 480 milliseconds;
  * Active or uncontrolled severe infection #≥ CTCAE level 2 infection#;
  * Known human immunodeficiency virus #HIV# infection; Known clinically significant history of liver disease, including viral hepatitis [known carriers of hepatitis B virus #HBV# must exclude active HBV infection, i.e. HBV DNA positivity #>1 × 104 copies/mL or>2000 IU/ml#; Known hepatitis C virus infection #HCV# and HCV RNA positivity #>1 × 103 copies/mL, or other types of hepatitis or cirrhosis;
  * According to the judgment of the researchers, patients deemed unsuitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  Overall Response Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastric Surgery， Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No